CLINICAL TRIAL: NCT00209417
Title: GEHC Has Decided Not to Provide This Detail But Will Rely on the Brief Title.
Brief Title: Renal Effects of Two Iodinated Contrast Media in Patients at Risk Undergoing Computed Tomography
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Supported by preliminary interim analysis. Not based on any safety signals in study or any quality issues that could affect efficacy of the product.
Sponsor: GE Healthcare (Industry)
Collaborators: ABX CRO (Other); Examination Management Services Inc. (Industry); Covance (Industry); Quintiles, Inc. (Industry); Averion International Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: DXV406
Record Dates: First submitted 2005-08-24; First posted 2005-09-21 (Estimated); Results first posted 2014-10-10 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Renal Insufficiency; Diabetes Mellitus
Keywords: Iodixanol; Iopamidol; computed tomography; Patients with pre-existing renal impairment and diabetes
MeSH Terms: conditions — Renal Insufficiency; Diabetes Mellitus | interventions — iodixanol; Iopamidol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Iodixanol 320-Arm 1 (Active Comparator): Iodixanol 320 mg I/mL
  Interventions: Drug: Iodixanol 320-Arm 1
- Iopamidol 300-Arm 2 (Active Comparator): Iopamidol 300 mg I/mL
  Interventions: Drug: Iopamidol 300-Arm 2

INTERVENTIONS:
Drug: Iodixanol 320-Arm 1
  Other Names: Visipaque
  Arms: Iodixanol 320-Arm 1
Drug: Iopamidol 300-Arm 2
  Other Names: Isovue
  Arms: Iopamidol 300-Arm 2

SUMMARY:
It is well known that X-ray contrast media can affect kidney function in some patients, especially when administered intra-arterially, and patients who already suffer from reduced kidney function and diabetes mellitus may be at increased risk. It is widely accepted to use low-osmolar or iso-osmolar contrast media, especially in patients at risk for contrast media-induced nephropathy. However, little is known about the intravenous use of X-ray contrast media in risk patients, such as contrast-enhanced CT examinations. The main purpose of this study is to evaluate and compare the effects on kidney function of two contrast media, the iso-osmolar iodixanol and the low-osmolar iopamidol in patients at risk of kidney damage associated with the injection of contrast media. Due to the iso-osmolar feature, it is expected less influence on renal function following administration of iodixanol. A standard hydration procedure, based on available guidelines will be given to all patients to prevent negative effects on the kidneys. Serum creatinine (SCr ) concentrations will be measured before and up to 7 days after contrast media administration to evaluate the effects on renal function.

DETAILED DESCRIPTION:
GEHC has decided not to provide this detail

ELIGIBILITY:
Inclusion Criteria:

* Patients with a combination of diabetes mellitus (type I or II) and renal impairment who are referred for a contrast-enhanced CT examination.

Exclusion Criteria:

* Concurrent administration of potentially nephroprotective or nephrotoxic drugs is not permitted.
* Patients undergoing dialysis or kidney transplantation will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Actual)
Dates: Start 2005-06; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Johnson, MS, MBA, Study Director — GE Healthcare
Locations (2):
- GE Healthcare, Princeton, New Jersey, United States
- GE Healthcare, Amersham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 656 subjects enrolled. 8 subjects did not continue on in the study. 7 of the 8 subjects discontinued the study prior to contrast media administration and 1 of the 8 subjects received a contrast media of unknown type and was excluded from the study.
  Subtracting 8 subjects from the total 656, a total of 648 subjects actually completed the study.
Groups:
- Iodixanol 320-Arm 1: Iodixanol 320 mg I/mL
  Iodixanol 320-Arm 1
- Iopamidol 300-Arm 2: Iopamidol 300 mg I/mL
  Iopamidol 300-Arm 2
Period: Overall Study
Arm/Group | Iodixanol 320-Arm 1 | Iopamidol 300-Arm 2
Started | 321 | 327
Completed | 321 | 327
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iodixanol 320-Arm 1 | Iopamidol 300-Arm 2 | Total
Number analyzed (Participants) | 321 | 327 | 648
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (12.02) | 66.5 (12.01) | 66.4 (12.01)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 133 | 136 | 269
  >=65 years | 188 | 191 | 379
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 170 | 317
  Male | 174 | 157 | 331
Region of Enrollment [Number; unit: participants]
  United States | 71 | 70 | 141
  United Kingdom | 10 | 14 | 24
  Austria | 11 | 12 | 23
  China | 45 | 48 | 93
  Czech Republic | 1 | 1 | 2
  France | 8 | 9 | 17
  Germany | 34 | 38 | 72
  Hungary | 6 | 8 | 14
  Italy | 4 | 5 | 9
  Poland | 60 | 55 | 115
  Russian Federation | 57 | 56 | 113
  Spain | 5 | 1 | 6
  Sweden | 6 | 8 | 14
  Switzerland | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Incidence Rate of Contrast Medium-Induced Nephropathy (CIN) Between Iodixanol and Iopamidol in Patients With Impaired Renal Function.
Description: The primary endpoint was the incidence rate of CIN, defined as an intra-individual increase in serum creatinine (SCr) of greater than or equal to 44.2 µmol/L (greater than or equal to 0.5 mg/dL).
  Subjects with a pre-contrast (baseline) serum creatinine value greater than or equal to 1.5 mg/dL for males and greater than or equal to 1.3 mg/dL for females or eGFR of less than or equal to 50 mL/min/1.73m squared, and a post-contrast serum creatinine value available on days 2 or 3, administered greater than or equal to100 mL or greater than or equal to 1.5 mL/kg bodyweight IMP, without presence of any major protocol violations, and without evidence of other causes inducing acute renal dysfunction.
Time Frame: From baseline up to 3 days post contrast administration.
Population: To calculate the incidence rate of CIN, divide the number of subjects affected by the total number of subjects dosed in each treatment group.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Iodixanol 320-Arm 1 | Iopamidol 300-Arm 2
Number analyzed (Participants) | 192 | 207
percentage of subjects | 9.90 [5.67 to 14.12] | 10.63 [6.43 to 14.83]

2. Secondary Outcome: Assessment of Overall Image Quality Between Iodixanol and Iopamidol in Patients Undergoing Contrast-enhanced Multi-detector-row Helical Computed Tomography (MDCT) Examination.
Description: Overall Image Quality rated as "Excellent, Good, Sufficient or Insufficient Poor" by radiologists blinded to the contrast administration.
Time Frame: Within 2, 3 and 7 days post contrast administration.
Measure: Number; unit: Number of images
Units Other Than Participants: Images Analyzed
Arm/Group | Iodixanol 320-Arm 1 | Iopamidol 300-Arm 2
Number analyzed (Participants) | 321 | 327
Number analyzed (Images Analyzed) | 321 | 327
Number of images
  Image Quality-Excellent | 220 | 207
  Image Quality-Good | 81 | 103
  Image Quality-Sufficient | 13 | 9
  Image Quality-Insufficient | 7 | 8

ADVERSE EVENTS:
Arm/Group | Iodixanol 320-Arm 1 | Iopamidol 300-Arm 2
Serious Adverse Events (participants affected / at risk) | 6/321 | 6/327
Other Adverse Events (participants affected / at risk) | 0/321 | 0/327
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iodixanol 320-Arm 1 (N=321) | Iopamidol 300-Arm 2 (N=327)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Renal failure Acute (Renal and urinary disorders) | 1 (1) | 1 (1) — Outcome was death for both Iodixanol and Iopamidol.
Renal Impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Outcome was death for Iodixanol.
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Outcome was death for Iodixanol.
Sudden Death (Cardiac disorders) | 0 (0) | 1 (1) — Outcome was death for Iopamidol.
Aortic Dissection (Cardiac disorders) | 0 (0) | 1 (1) — Outcome was death for Iopamidol.
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blood Lactic Acid Increase (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Coma (Vascular disorders) | 0 (0) | 1 (1)
Sepsis (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1) — Outcome was death for Iopamidol.
Cerebrovascular Accident (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No